CLINICAL TRIAL: NCT04485117
Title: Propofol Versus Sevoflurane Anesthesia in Pediatric Strabismus Surgery: Feasibility of BIS Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIS Monitoring in Strabismus
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Strabismus
Keywords: Bispectral Index Monitoring
MeSH Terms: conditions — Strabismus | interventions — Consciousness Monitors; Laryngeal Masks; Sevoflurane; Propofol; Anesthesia, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Group (Active Comparator): Laryngeal mask airway is inserted and anesthesia is maintained with sevoflurane anesthesia under BIS monitoring.
  Interventions: Device: Bispectral Index Monitor; Device: Laryngeal Mask Airway; Drug: Sevoflurane
- Propofol Group (Active Comparator): Laryngeal mask airway is inserted and anesthesia is maintained with propofol infusion under BIS monitoring.
  Interventions: Device: Bispectral Index Monitor; Device: Laryngeal Mask Airway; Drug: Propofol

INTERVENTIONS:
Device: Bispectral Index Monitor — Bispectral Index (BIS) sensor electrodes are applied over the patient's forehead after cleaning the forehead thoroughly with an alcohol swab.
  Other Names: BIS Monitoring
Device: Laryngeal Mask Airway — Capnography connected to laryngeal mask airway is introduced after adequate jaw relaxation and oral airway tolerance; its size is chosen according to the body weight of the child.
  Other Names: Supraglottic Airway Device
Drug: Sevoflurane — Anesthesia is induced inhalationally by face mask with 8% sevoflurane in 100% oxygen, then decreased to 2-3% in 40% oxygen thoroughout the operation for maintenance of anesthesia.
  Other Names: Inhalational Anesthesia
  Arms: Sevoflurane Group
Drug: Propofol — Anesthesia is induced by propofol (2mg/kg), then maintained using an infusion of fixed concentration (10-15 mg/kg/h) as titrated by the anesthesiologist .
  Other Names: Intravenous Anesthesia
  Arms: Propofol Group

SUMMARY:
This study is conducted to evaluate importance of bispectral index (BIS) monitoring in patients undergoing strabismus surgery when using propofol in comparison to sevoflurane anesthesia regarding their effects on oculocardiac reflex, intraoperative hemodynamic stability, emergence agitation, postoperative pain, nausea and vomiting.

DETAILED DESCRIPTION:
Strabismus surgery can cause unfavorable side effects during intraoperative and postoperative periods including increased risk of the oculocardiac reflex, hemodynamic instability, emergence agitation, postoperative pain, nausea and vomiting. Sevoflurane is an inhalation anesthetic widely used in pediatric anesthesia with minimal airway irritation. Propofol is an intravenous sedative-hypnotic agent with amnestic properties that causes loss of consciousness. Bispectral index monitor provide some more evidence that deeper anesthesia can provide some protection against the oculocardiac reflex. Therefore, this study is conducted to evaluate the role of BIS monitoring in comparing the use of propofol and sevoflurane anesthesia in pediatric strabismus surgery.

This prospective, randomized, comparative clinical study will include 100 children who are scheduled for elective strabismus surgery under general anesthesia in Mansoura ophthalmology center. Informed written consent is obtained from parents of all subjects in the study after ensuring confidentiality. The study protocol is explained to parents of all patients in the study who are kept fasting prior to surgery. Patients are randomly assigned to two equal groups according to computer-generated table of random numbers using the permuted block randomization method. The collected data are coded, processed, and analyzed using SPSS program. All data are considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for elective Strabismus surgery.

Exclusion Criteria:

* Parental refusal of consent.
* Hyperactive airway disease or respiratory diseases.
* Children with developmental delays, mental or neurological disorders.
* Bleeding or coagulation diathesis.
* History of known sensitivity to the used anesthetics.
* Children with previous surgery in the eye.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Incidence of oculocardiac reflex | Up to the end of the surgery
  Any dysrhythmia or rapid reduction in HR by more than 25% from the baseline is taken as oculocardiac reflex.

SECONDARY OUTCOMES:
Changes in bispectral index | Up to the end of the surgery
  Bispectral index values (0-100) are recorded every five minutes until the end of the surgery
Changes in heart rate | Up to the end of the surgery
  Heart rate (beat/min) is recorded at five-minute intervals until the end of the surgery
Changes in mean arterial blood pressure | Up to the end of the surgery
  Mean blood pressure (mmHg) is recorded at five-minute intervals until the end of the surgery
Changes in postoperative emergence agitation scale | Up to 30 minutes after surgery
  Agitation is assessed using the 5- step Cravero scale (1-5) every five minutes from awakening and for 30 minutes.(1:Obtunded with no response to stimulation, 2:Asleep but responsive to movement or stimulation, 3:Awake and responsive, 4:Crying, 5:Thrashing behaviour that requires restraint)
Changes in postoperative pain score | Up to 24 hours after surgery
  Pain score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) is assessed every two hours for 24 hours after surgery.
First analgesic request | Up to 24 hours after surgery
  The time of the first analgesic request for paracetamol is recorded.
Total analgesic requirements of paracetamol | Up to 24 hours after surgery
  The amount of paracetamol consumption given as a rescue analgesia to patients is measured all over the 24 hours.
Incidence of postoperative nausea and vomiting | Up to 24 hours after surgery
  Incidence of postoperative nausea and vomiting is assessed during the first 24 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No